CLINICAL TRIAL: NCT01609400
Title: An Extension of CTN 31GB0607 to Evaluate Long Term Safety of NASHA Treatment in the Breast
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 31GB1103
Record Dates: First submitted 2012-05-08; First posted 2012-06-01 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2015-02

CONDITIONS: Breast Enhancement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast enhancement

SUMMARY:
The study evaluates degradation of NASHA in breast 4 and 6 years post treatment, long term safety and evaluation if a satisfactory breast cancer screening can be performed in subjects treated with NASHA-gel in breast. An independent evaluation of the aesthetic changes is also performed.

ELIGIBILITY:
Inclusion Criteria:

* subject treated with NASHA-gel in the breasts in study 31GB0607
* signed informed consent

Exclusion Criteria:

* no exclusion criteria in this study

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects treated in study 31GB0607
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluate if study product has been completely degraded in the breast 4 years post treatment in study 31GB0607, using MRI | 4 years
Evaluate if study product has been completely degraded in the breast 6 years post treatment in study 31GB0607, using MRI | 6 years

SECONDARY OUTCOMES:
Evaluate long term safety of study product in breast enhancement using adverse events reporting, breast examination, ultrasound and mammography. | 4 years
Perform an independent evaluation of aesthetic changes in the treated breasts taking into consideration the aging of the subject, using pre- and post-treatment photos | 4 years
Evaluate if a satisfactory breast cancer screening can be performed in subjects treated with NASHA-gel in breast(s) | 4 years
Evaluate long term safety of study product in breast enhancement using adverse events reporting, breast examination, ultrasound and mammography. | 6 years
Perform an independent evaluation of aesthetic changes in the treated breasts taking into consideration the aging of the subject, using pre- and post-treatment photos | 6 years
Evaluate if a satisfactory breast cancer screening can be performed in subjects treated with NASHA-gel in breast(s) | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, M.D., Principal Investigator — Akademikliniken, Stockholm, Sweden; Michael Olenius, M.D., Principal Investigator — Proforma Clinic AB, Stockholm, Sweden